CLINICAL TRIAL: NCT04593784
Title: A Phase 2 Randomized, Double-blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Ciraparantag for Reversal of Anticoagulation in Healthy Adults
Brief Title: Study of Ciraparantag for Reversal of Anticoagulation Induced by Edoxaban, Apixaban or Rivaroxaban in Healthy Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision unrelated to safety
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Ciraparantag Holdings GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AMAG-977-213
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: ciraparantag; PER977; Apixaban; Rivaroxaban; Whole Blood Clotting Time (WBCT); Coagulometer; AMAG 977; Edoxaban
MeSH Terms: interventions — PER977

STUDY DESIGN:
Intervention Model Description: The study will be conducted in separate cohorts; each cohort will evaluate the reversal of a different anticoagulant drug. Within each cohort, an initial group of subjects (Group 1) will be enrolled for evaluation of a target dose of ciraparantag. Depending on the efficacy and safety results from Group 1, a second group (Group 2) may be enrolled to evaluate a different dose of ciraparantag for that cohort.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Anticoagulant drugs will be administered in an open-label manner. Ciraparantag or placebo (PBO) will be administered in a double-blind manner. Subjects and all study site personnel except the study pharmacist will be blinded to individual subject treatment assignment (ciraparantag or PBO). The Sponsor will be unblinded to individual treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Subjects receive 60 mg edoxaban orally once daily in the morning on Days 1 to 4. On Day 4, approximately 3 hours after administering edoxaban, study drug (ciraparantag or placebo) will be intravenously administered.
  Interventions: Drug: Ciraparantag; Drug: Placebo; Device: Point-of-Care Coagulometer (investigational device)
- Cohort 2 (Experimental): Subjects receive 10 mg apixaban orally every 12 hours on Days 1 to 3, with a final dose in the morning on Day 4. On Day 4, approximately 4 hours after administering apixaban, study drug (ciraparantag or placebo) will be intravenously administered.
  Interventions: Drug: Ciraparantag; Drug: Placebo; Device: Point-of-Care Coagulometer (investigational device)
- Cohort 3 (Experimental): Subjects receive 20 mg rivaroxaban orally once daily in the morning on Days 1 to 4. On Day 4, approximately 4 hours after administering rivaroxaban, study drug (ciraparantag or placebo) will be intravenously administered.
  Interventions: Drug: Ciraparantag; Drug: Placebo; Device: Point-of-Care Coagulometer (investigational device)

INTERVENTIONS:
Drug: Ciraparantag — Ciraparantag: 180 mg, intravenous
  Other Names: PER977; AMAG 977
Drug: Placebo — Placebo: 0.9% sodium chloride, intravenous
  Other Names: PBO
Device: Point-of-Care Coagulometer (investigational device) — Perosphere Technologies' Point of Care (POC) Coagulometer Device will be used to measure whole blood clotting time.
  Other Names: Coagulometer

SUMMARY:
A randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of ciraparantag for reversal of anticoagulation induced by different anticoagulant drugs in generally healthy adults as measured primarily by an automated coagulometer device.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of ciraparantag for reversal of anticoagulation induced by different anticoagulant drugs (edoxaban, apixaban or rivaroxaban) in generally healthy adults. Throughout the study, coagulation status will be determined by whole blood clotting time (WBCT), which will be measured primarily by the Perosphere Technologies' PoC Coagulometer and at selected timepoints using a manual testing method.

The study will be conducted in three separate cohorts; each cohort will evaluate the reversal of a different anticoagulant drug. Within each cohort, an initial group of subjects (Group 1) will be enrolled for evaluation of a target dose of ciraparantag. Depending on the efficacy and safety results from Group 1, a second group (Group 2) may be enrolled to evaluate a different dose of ciraparantag for that cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. 18 to 75 years of age.
3. Be in generally good health
4. BMI 18 to 32 kg/m2, inclusive, at Screening.
5. If female, be surgically sterile or post-menopausal or if of child-bearing potential, using an acceptable method of contraception (other than a combination estrogen/progestin hormonal contraceptive) for at least 1 month prior to Day 1.
6. If male, be surgically sterile, or agree to use appropriate contraception.
7. Have suitable venous access for multiple venipunctures.

Exclusion Criteria:

1. Have any of the following findings at Screening:

   1. Hemoglobin or hematocrit value outside the normal range
   2. Platelet count outside the normal range
   3. PT or aPTT outside the normal range
   4. Plasma fibrinogen outside the normal range
   5. Serum triglycerides or total cholesterol outside the normal range
   6. Serum creatinine >1.5 mg/dL (133 μmol/L) or known renal disease
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x the upper limit of normal, or known liver disease
   8. Total bilirubin outside the normal range
   9. Positive viral screen for hepatitis B virus, hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
   10. Positive pregnancy test (females)
   11. Positive drug, tobacco or alcohol screen
   12. Any clinically significant findings on 12-lead ECG or urinalysis
2. Have a personal or family history of clotting disorder or hematologic abnormality.
3. Have a history of unexplained syncope.
4. Have a history within 6 months prior to Screening of major bleeding, trauma, surgical procedure of any type, or vaginal delivery
5. Have a history within 6 months prior to Screening of peptic ulcer or gastrointestinal bleeding.
6. Have received any blood product or anticoagulant within 3 months prior to Screening.
7. Have donated blood or blood products within 3 months prior to Screening
8. Have a history of minor bleeding episodes within 1 month prior to Screening, or a long-standing history of such bleeding.
9. If female, have a history of excessive or dysfunctional uterine bleeding (unless the subject had a subsequent hysterectomy).
10. Have used any tobacco or nicotine-containing products within 3 months prior to Screening.
11. Have used any systemic prescription or non-prescription drugs within 14 days prior to Day 1 (except for permitted contraceptives).
12. If female, be pregnant, breastfeeding, or planning to become pregnant during the study.
13. Have received ciraparantag in any prior clinical study.
14. Have received another investigational drug within 5 half-lives or 30 days, whichever is longer, prior to Day 1.
15. Known allergy to edoxaban, apixaban or rivaroxaban.
16. Have any other condition that, in the opinion of the Investigator, would interfere with a subject's ability to adhere to the protocol, interfere with assessment of the investigational product, or compromise the safety of the subject or the quality of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
The number of subjects achieving WBCT ≤120% of baseline within 1 hour after administration of ciraparantag or placebo and sustained after 1 hour through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours

SECONDARY OUTCOMES:
The number of subjects achieving WBCT ≤115% of baseline within 1 hour after administration of ciraparantag or placebo and sustained after 1 hour through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤110% of baseline within 1 hour after administration of ciraparantag or placebo and sustained after 1 hour through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤120% of baseline within 30 minutes after administration of ciraparantag or placebo and sustained after 30 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤115% of baseline within 30 minutes after administration of ciraparantag or placebo and sustained after 30 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤110% of baseline within 30 minutes after administration of ciraparantag or placebo and sustained after 30 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤120% of baseline within 15 minutes after administration of ciraparantag or placebo and sustained after 15 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤115% of baseline within 15 minutes after administration of ciraparantag or placebo and sustained after 15 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
The number of subjects achieving WBCT ≤110% of baseline within 15 minutes after administration of ciraparantag or placebo and sustained after 15 minutes through at least 6 hours after ciraparantag/placebo dosing. | 6 Hours
Correlation between WBCT measured with Perosphere Technologies' POC Coagulometer and with a manual testing method | 24 Hours
  Correlation will be analyzed by a linear regression model.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Qps-Mra, Llc., South Miami, Florida
  - Frontage Clinical Services, Secaucus, New Jersey
  - ICON Early Phase Services, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No